CLINICAL TRIAL: NCT00876785
Title: Effect of Rye Bread Breakfasts on Subjective Hunger and Satiety
Brief Title: Effect of Rye Bread Breakfasts on Eight Hour Satiety Ratings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Lantmännen R&D (Unknown); Good Food Practice, Sweden (Industry)
Responsible Party: Hanna Isaksson, lantmännen R&D
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SI829
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: Rye bread satiety breakfast
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Reference wheat bread breakfast
  Interventions: Other: wheat bread based breakfast
- 2 (Experimental): Rye bread breakfast
  Interventions: Other: Rye bread breakfast

INTERVENTIONS:
Other: Rye bread breakfast — A randomised, within-subject comparison design was used. Appetite (hunger, satiety and desire to eat) was rated regularly from just before breakfast at 08:00 until 16:00. Amount, type and timing of food and drink intake during the study period were standardised.
  Arms: 2
Other: wheat bread based breakfast — Reference wheat bread breakfast
  Arms: 1

SUMMARY:
The aim of the present study was to investigate subjective appetite during 8 hours after intake of iso-caloric rye bread breakfasts varying in dietary fiber composition and content.

DETAILED DESCRIPTION:
Energy-dense foods that require little effort to consume and that are rapidly digested may cause passive over-consumption by failure to provide a feeling of fullness corresponding to the energy content. A diet that is predominantly based on such foods may lead to overweight. It is therefore important to identify properties of foods that facilitate energy balance by creating a high satiety per calorie. A number of studies have confirmed that foods naturally rich in dietary fiber promote the feeling of fullness and reduce hunger in the short term.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 60 years
* body mass index (BMI) 18-27 kg/m2
* a habit of consuming breakfast, lunch and dinner everyday
* fasting plasma glucose 4.0-6.1 mmol/L
* haemoglobin (Hb) in men 130-170 g/L, in women 120-150 g/L
* thyroid-stimulating hormone (TSH) 0.3-4.0 mlE/L
* willingness to comply with the study procedures

Exclusion Criteria:

* intake of medicine likely to affect appetite or food intake
* any medical condition involving the gastrointestinal tract
* eating disorder
* smoking
* consumption of more than three cups of coffee per day
* change in body weight of more than 10% three months prior to screening
* consumption of any restricted diet such as vegan, gluten-free, slimming etc.
* pregnancy, lactation or wish to become pregnant during the study period

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Subjective satiety, hunger and desire to eat | During 8 hours after intake of test meal

CONTACTS AND LOCATIONS:
Overall Officials: Per Aman, Professor, Study Director — university
Locations (1):
- Swedish University of Agricultural Sciences, Uppsala, Sweden

REFERENCES:
- [Derived] Isaksson H, Fredriksson H, Andersson R, Olsson J, Aman P. Effect of rye bread breakfasts on subjective hunger and satiety: a randomized controlled trial. Nutr J. 2009 Aug 26;8:39. doi: 10.1186/1475-2891-8-39. PMID 19709412